CLINICAL TRIAL: NCT02934555
Title: Ubiquinol as a Metabolic Resuscitator in Post-Cardiac Arrest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Principal Investigator, Michael Donnino, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2015P000319
Record Dates: First submitted 2016-01-18; First posted 2016-10-17 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — ubiquinol; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Patients in the control group will receive a liquid placebo, which is 50 mL of Ensure (a dietary supplement). This will be given every 12 hours for 7 days, until neurologic recovery, or until hospital discharge.
  Interventions: Dietary Supplement: Ensure
- Ubiquinol (Experimental): Patients in the experimental group will receive 300 mg of Ubiquinol in a liquid mixture. The liquid Ubiquinol will be mixed with 50 mL of Ensure (a dietary supplement) to ensure blinding. This will be given every 12 hours for 7 days, until neurologic recovery, or until hospital discharge.
  Interventions: Drug: Ubiquinol; Dietary Supplement: Ensure

INTERVENTIONS:
Drug: Ubiquinol — 300 mg Ubiquinol (3 mL liquid Ubiquinol).
  Other Names: CoQ10
  Arms: Ubiquinol
Dietary Supplement: Ensure — 50 mL Ensure

SUMMARY:
To study the effects of ubiquinol as a "metabolic resuscitator" in post-cardiac arrest.

DETAILED DESCRIPTION:
Cardiac arrest (CA) occurs in more than 400,000 patients in the United States each year with an estimated mortality of greater than 90%. The majority of patients who are resuscitated from CA will succumb to the neurologic morbidity associated with the post-CA syndrome and ischemic-reperfusion injury. Currently, there are no pharmacologic agents known to offer survival benefit or to prevent devastating neurologic injury in post-CA patients.

A potential therapeutic target following ischemia-reperfusion injury is mitochondrial function in the injured cell and/or reduction of oxygen free radicals. Coenzyme Q10 (CoQ10) is an essential mitochondrial co-factor and free radical scavenger that has been proposed as a neuroprotective agent in various neurodegenerative disorders as well as a cardioprotective agent. CoQ10 have furthermore shown exciting preliminary results as a potential therapy in post-CA.

In order to test the effects of ubiquinol as a "metabolic resuscitator" in post-CA patients and to provide additional preliminary data for a large-scale clinical trial, the investigators are conducting a randomized, double-blind, place-controlled trial of ubiquinol in post-CA patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Cardiac arrest defined by cessation of pulse requiring chest compressions
* Not following commands after ROSC
* Admission to the ICU
* Naso/orogastric tube
* Ability to receive enteral medication

Exclusion Criteria:

* Protected populations (pregnant women, prisoners, the intellectual disabled)
* Current CoQ10 supplementation
* Anticipated death within 24 hours
* > 12 hours from ROSC to estimated randomization
* Jejunostomy tube (J-tube)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05-25 (Actual); Study Completion 2019-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 50 mL of Ensure (a dietary supplement) every 12 hours for 7 days, until neurologic recovery, or until hospital discharge.
- Ubiquinol: 300 mg of Ubiquinol mixed with 50 mL of Ensure (a dietary supplement) every 12 hours for 7 days, until neurologic recovery, or until hospital discharge.
Period: Overall Study
Arm/Group | Placebo | Ubiquinol
Started | 23 | 25
Completed (Endpoint measurements available) | 21 | 22
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ubiquinol | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [57 to 79] | 60 [46 to 69] | 62 [52 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 16 | 18 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 6 | 18
  Other | 11 | 19 | 30
Number of Participants with Shock [Count of Participants; unit: Participants]
  Shock | 14 | 16 | 30
  Non-shock | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Coenzyme Q10 Plasma Levels
Description: Total (oxidized and reduced form) coenzyme Q10
Time Frame: Up to 72 hours
Population: Blood samples were not available on all participants at all time-points.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 23 | 25
ng/mL
  0 hours: number analyzed (Participants) | 22 | 25
  0 hours | 185 [120 to 267] | 207 [125 to 348]
  24 hours: number analyzed (Participants) | 21 | 20
  24 hours | 113 [94 to 208] | 441 [215 to 510]
  48 hours: number analyzed (Participants) | 15 | 18
  48 hours | 148 [85 to 299] | 615 [286 to 817]
  72 hours: number analyzed (Participants) | 13 | 16
  72 hours | 157 [102 to 169] | 554 [380 to 1200]

2. Secondary Outcome: Decreased Neurological Injury
Description: Neuron Specific Enolase levels
Time Frame: Up to 72 hours
Population: Blood samples were not available on all participants at all time-points.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 23 | 25
ng/mL
  0 hours: number analyzed (Participants) | 22 | 24
  0 hours | 7.6 [5.9 to 10.7] | 9.2 [6.7 to 14.3]
  24 hours: number analyzed (Participants) | 21 | 21
  24 hours | 8.2 [4.3 to 19.1] | 16.8 [9.5 to 19.8]
  48 hours: number analyzed (Participants) | 16 | 19
  48 hours | 5.3 [2.9 to 9.2] | 12.6 [4.3 to 22.6]
  72 hours: number analyzed (Participants) | 14 | 17
  72 hours | 6.8 [4.0 to 14.4] | 14.4 [4.0 to 18.4]

3. Secondary Outcome: Cellular Oxygen Consumption
Description: Cellular (peripheral blood mononuclear cells) oxygen consumption measured with the XFe24 Extracellular Flux Analyzer
Time Frame: At 24 hours
Population: Cellular oxygen consumption was measured in a subset of the total cohort.
Measure: Median (Inter-Quartile Range); unit: mL/min/mg
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 21 | 22
mL/min/mg
  Basal OCR | 7.6 [5.5 to 9.0] | 6.5 [3.7 to 9.3]
  Maximal OCR | 20.7 [16.1 to 34.5] | 18.0 [10.8 to 32.0]

4. Secondary Outcome: Global Oxygen Consumption
Description: VO2 measured using a Compact Anesthesia monitor
Time Frame: Up to 48 hours
Population: Global oxygen consumption was measured in a subset of the total cohort.
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 18 | 14
mL/min/kg
  12 hours | 3.1 [2.6 to 3.9] | 3.5 [3.0 to 3.9]
  24 hours | 3.2 [3.0 to 3.6] | 3.5 [2.9 to 4.5]
  48 hours | 3.8 [2.9 to 4.8] | 4.4 [3.9 to 5.3]

5. Secondary Outcome: Mortality
Description: In-hospital mortality
Time Frame: At hospital discharge, an average of 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 23 | 25
Participants | 14 | 15

6. Secondary Outcome: Number of Participants With Favorable Neurological Outcome
Description: Favorable Neurological Outcome as measured by the Cerebral Performance Category (CPC 1-2) score. A CPC score of 1 (mild or no neurological deficit) or 2 (moderate disability) was defined as a favorable neurological outcome. A CPC score of 3 (severe disability), 4 (vegetative state), or 5 (death) was defined as an unfavourable neurological outcome.
Time Frame: At hospital discharge, an average of 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 23 | 25
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: From enrolment until hospital discharge.
Arm/Group | Placebo | Ubiquinol
All-Cause Mortality (participants affected / at risk) | 14/23 | 15/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02934555/Prot_SAP_000.pdf